CLINICAL TRIAL: NCT05647759
Title: Rural HEART Camp Connect: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0773-20-FB
Record Dates: First submitted 2022-11-11; First posted 2022-12-12 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
Keywords: cardiac rehabilitation; exercise adherence; virtual coaching
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-group, repeated measures feasibility study.
Masking Description: If consent is obtained in person, study personnel will be in a private room with both parties masked, eye protection, and social distancing guidelines in place. Baseline data collection will occur in a private room with masks, eye protection, and social distancing guidelines in place. Hospital-based facilities and staff are in compliance with local health department guidance on masks and social distancing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEART Camp Connect (Experimental): Participants will have access to a virtual exercise platform or membership to a medical exercise facility. Participants will meet with a virtual exercise coach via zoom on a weekly basis.
  Interventions: Behavioral: HEART Camp Connect

INTERVENTIONS:
Behavioral: HEART Camp Connect — Once eligible and enrolled, participants will aim to complete 150 minutes of moderate-intensity exercise a week with the help of a virtual exercise coach

SUMMARY:
This study builds on the tested and refined HEART Camp intervention which has been shown to improve long-term adherence to exercise in individuals diagnosed with heart failure. HEART Camp Connect enhances HEART Camp by delivering the coaching via videoconference and providing access to hospital-based exercise facilities and online exercise programming. This study is a prospective, single-group, repeated measures feasibility study with 4 data collection points (baseline, 4, 8, and 12 weeks). Study variables including instruments will be collected at baseline, 4, and 8 weeks. Participants will also be asked to participate in a 30-45 minute interview at 12 weeks.

DETAILED DESCRIPTION:
At a rural health center in central Nebraska, potential participants will be identified, screened, and approached for participation. Study personnel will obtain informed consent in person in a private room or over the phone facilitated by the University of Nebraska Medical Center (UNMC) electronic consent process. Once consented, participants will complete cardiopulmonary exercise testing (CPET) to guide individual exercise prescriptions and protect against risks associated with exercise. CPET results that preclude safe exercise training (arrhythmia) or those with CPET results indicating cardio-respiratory fitness (females with maximum oxygen consumption ≥ 21ml/kg/min and males with oxygen consumption ≥ 24 ml/kg/min) will be withdrawn from the study.

Study personnel will complete baseline data collection (demographics, survey collection, and 6-minute-walk-test) on all participants at enrollment. The survey instruments have been validated and will be repeated at weeks 4 and 8. Participants will be given instruction on the use of the Actigraph, Polar Watch and chest strap, and Activity/Exercise Diary. The Actigraph will be worn for 7 consecutive days at baseline, week 4, and week 8. Participants will be asked to record daily activity/exercise in their diary for the entirety of the 12-week study and will be shared weekly with their coach. Participants will wear their Polar Watch and chest strap during exercise sessions for heart rate monitoring.

Prior to beginning exercise on their own, participants will complete 6 supervised, monitored sessions in cardiac rehabilitation. During these sessions, participants will be monitored by cardiac rehabilitation staff for adverse events during moderate-intensity aerobic exercise (40-80% of heart rate reserve) and resistance training (10-15 repetitions to volitional fatigue). During these sessions, participants will also receive educational training via videos on topics such as exercising with heart failure, how medications impact exercise, and nutrition. If a participant does not complete the sessions or is deemed unsafe to exercise, he/she will not be eligible to continue in the study.

Participants will be instructed to wear a heart rate monitor (Polar Watch and chest strap) during all exercise sessions and strive to meet a goal of 150 minutes of moderate-intensity exercise per week. Minutes toward adherence goals for the study will be calculated as time spent participating in a moderate-intensity activity and determined by their CPET results and personalized exercise prescription. Participants will be familiar with using heart rate and Rating of Perceived Exertion (RPE) to guide their exercise from their participation in the 6 supervised sessions. The heart rate monitor will be blue-tooth enabled and will require connection to the internet.

Participants will be given the choice to exercise at a hospital-based exercise facility, at home, or as a hybrid approach. If exercising at home, participants will be provided with training plans that will be available online or in hard-copy forms.

Each participant will be given access to an Omaha-based exercise coach that he/she will meet with weekly over Zoom for 30 minutes. Coaches will discuss exercise over the past week including problems, issues, concerns. Goals will be set, reviewed, assessed, and revised each week.

All participants will be given paid access to a hospital-based fitness facility for 8 weeks out of this 12-week study. Weeks 9-12 of the study, participants may elect to self-pay for membership or exercise at home. Exercise diaries will continue to be collected and Polar watch data will be monitored by exercise coaches until the end of this 12-week study. Participants will not meet with their exercise coach during the final 4 weeks. The rationale for this is that ultimately our goal is for participants to develop self-efficacy, knowledge, and positive attitudes toward exercise that will allow them to adhere to exercise without our intervention. The hope is that 8 weeks of exercise training and weekly coaching will get them started and they will continue on their own after that.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure with preserved ejection fraction or heart failure (HF) with reduced ejection fraction (Stage C, chronic HF confirmed by echocardiography and clinical evaluation)
* 19 years of age or older
* Stable pharmacologic therapy per guidelines for preceding 30 days
* Able to read and understand English.

Exclusion Criteria:

* Clinical evidence of decompensated heart failure
* Unstable angina
* Myocardial infarction, coronary artery bypass surgery, or biventricular pacemaker less than 6 weeks prior
* Orthopedic or neuromuscular disorders preventing participating in aerobic exercise
* Pregnancy
* Participation in 3 times per week aerobic exercise during the past 6 months
* Plans to move more than 50 miles from the exercise facility in the next 12 weeks
* Cardiopulmonary stress test results that preclude safe exercise training (arrhythmia) or cardiorespiratory fitness indicated by females with maximum oxygen consumption ≥ 21ml/kg/min and males with maximum oxygen consumption ≥ 24 ml/kg/min.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of administering Rural HEART Camp Connect | Baseline
  Feasibility of administering an exercise intervention with the help of virtual exercise coaches to rural patients with heart failure including assessments of process, resources, and procedures as described below.
  Process Recruitment and retention monitoring, records of participant attendance at all sessions, monitor minutes coached for all HEART Camp participants
  Resources - staff availability, accessibility, staff training
  Procedures Identify connectivity issues, the number of potential participants without smart devices with optimal capacity for the HEART Camp Connect, and evaluating orientation to the Polar watch, rating of perceived exertion and digital diaries
  Data Management Ease of data collection including time to complete instruments, technological transfer of data, and patterns of missing data on an ongoing basis
Determine perceptions of Rural HEART Camp connect in study participants | 12 weeks
  Qualitative interviews will explore perceptions of all study procedures, including use of home-based exercise and virtual coaching.

CONTACTS AND LOCATIONS:
Overall Officials: Windy W Alonso, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States